CLINICAL TRIAL: NCT06409871
Title: Impact of Methylxanthine Intake and Blue Light Exposure on Adhesive Shoulder Capsulitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, RAFAEL GUZMAN GARCIA, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Adhesive shoulder capsulitis
Record Dates: First submitted 2024-05-02; First posted 2024-05-10 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Adhesive Capsulitis of Shoulder
Keywords: Adhesive Shoulder Capsulitis; Metabolic Profile; Inflammation Mediators; Insomnia Disorders; Biological Rhythms
MeSH Terms: conditions — Bursitis; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy treatment (Placebo Comparator): Conventional physiotherapy treatment will be applied. The duration will be two weekly sessions of about 50 minutes, for 6 weeks.
  Interventions: Other: Physiotherapy treatment.
- Physiotherapy treatment and modification of the biorhythm (Experimental): The same physiotherapy treatment will be applied together with the modification of their biorhythm. This will be recorded in a diary for 6 weeks, in which the time of going to bed and waking up will be recorded, together with the observation of the change in biorhythm. This group will also be provided with a second informed consent form including a data collection commitment document. The duration will be two weekly sessions of about 50 minutes, for 6 weeks.
  Interventions: Other: Physiotherapy treatment and modification of the biorhythm.

INTERVENTIONS:
Other: Physiotherapy treatment. — -Physiotherapy treatment will consist of joint mobilisation, proprioceptive neuromuscular facilitation and manual therapy.
  Arms: Physiotherapy treatment
Other: Physiotherapy treatment and modification of the biorhythm. — * Physiotherapy treatment will consist of joint mobilisation, proprioceptive neuromuscular facilitation and manual therapy.
  * Modification of the biorhythm will consist of eliminating methylxanthine-rich foods and/or beverages from their diet, as well as no exposure to electronic devices two hours before bedtime.
  Arms: Physiotherapy treatment and modification of the biorhythm

SUMMARY:
Adhesive shoulder capsulitis is a condition characterised by stiffness or lack of mobility of the shoulder. This results in a negative impact on quality of life and increased health care costs. Inflammation is a key factor in the pathogenesis of these patients. In addition, poor sleep quality and/or sleep deprivation can increase the production of pro-inflammatory cytokines, which contributes to the development of chronic inflammatory and metabolic diseases.

The most important function of sleep is recovery. Good sleep promotes healing, aids in the recovery of the immune, neurological, musculoskeletal systems and is necessary for pain sufferers to improve. The quantity and quality of sleep has an impact on the subject's inflammatory and metabolic markers.

In relation to the quantity and quality of sleep, it has been shown that foods and/or beverages rich in methylxanthine such as coffee, tea and chocolate can alter these parameters. As is the case with exposure to blue light emitted by electronic devices. The population are faced with deep-rooted habits in their daily lives that do not help to control pain in these patients.

HYPOTHESIS:

Due to the above, the following hypothesis is established:

Lack of consumption of food or beverages rich in methylxanthine and limiting the use of mobile devices two hours before going to sleep favours recovery from adhesive shoulder capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with adhesive shoulder capsulitis aged between 18 and 60 years.

Exclusion Criteria:

* Locked shoulder dislocations, shoulder arthritis, shoulder fractures, avascular necrosis, previous surgery in the hypochondrium region within the last year, having a medical or skin condition that prevents them from receiving tactile stimuli in the shoulder area, presence of a neurological or motor disorder, having diagnosed psychopathology, visual impairment, or subjects with other diseases that may affect sleep quality or inflammatory parameters.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Pain and Disability Questionnaire (SPADI) | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  It is a quality of life questionnaire developed to assess pain and disability associated with shoulder dysfunction. The SPADI is a 13-item shoulder function index of responders' ability to perform basic activities of daily living. Each item is scored using a numerical rating scale ranging from zero (no pain/no difficulty) to ten (worst pain imaginable/so difficult that help was required). SPADI provides a pain scale (five items; scale score range from zero to 50 points, expressed as a percentage) and a disability scale (eight items; scale score range from zero to 80 points, expressed as a percentage). The scores of the two scales are averaged to obtain a total Spanish version of the SPADI score (zero to 100 points). A higher score indicates greater pain-related disability.
Fasting glucose Metabolic Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  Fasting glucose (mg/dl) was measured. Blood sample was obtained following the guidelines of the National Biobank Network.
Insulin Metabolic Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  Insuline (mU/L) was measured. Blood sample was obtained following the guidelines of the National Biobank Network.
HOMA Index Metabolic Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  HOMA index was measured. Blood sample was obtained following the guidelines of the National Biobank Network.
Leptin Metabolic Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  Leptin (ng/ml) was measured. Blood sample was obtained following the guidelines of the National Biobank Network.
Triglycerides Metabolic Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  Triglycerides (mg/dl) was measured. Blood sample was obtained following the guidelines of the National Biobank Network.
Total Colesterol Metabolic Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  Total colesterol (mg/dl) was measured. Blood sample was obtained following the guidelines of the National Biobank Network.
HDL Colesterol Metabolic Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  HDL colesterol (mg/dl) was measured. Blood sample was obtained following the guidelines of the National Biobank Network.
Uric Acid Metabolic Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  Uric acid (mg/dl) was measured. Blood sample was obtained following the guidelines of the National Biobank Network.
High-sensitivity C-reactive Protein Metabolic Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  High-sensitivity C-reactive Protein (mg/L) was measured. Blood sample was obtained following the guidelines of the National Biobank Network.
IL-1 Inflammatory Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  IL-1 (pg/ml) was measured. The analysis of this inflammatory cytokines was conducted using ELISA (Enzyme-Linked Immunosorbent Assay), with a blood sample obtained according to the guidelines of the National Biobank Network.
IL-6 Inflammatory Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  IL-6 (pg/ml) was measured. The analysis of this inflammatory cytokines was conducted using ELISA (Enzyme-Linked Immunosorbent Assay), with a blood sample obtained according to the guidelines of the National Biobank Network.
IL-17 Inflammatory Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  IL-17 (pg/ml) was measured. The analysis of this inflammatory cytokines was conducted using ELISA (Enzyme-Linked Immunosorbent Assay), with a blood sample obtained according to the guidelines of the National Biobank Network.
IL-10 Inflammatory Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  IL-10 (pg/ml) was measured. The analysis of this inflammatory cytokines was conducted using ELISA (Enzyme-Linked Immunosorbent Assay), with a blood sample obtained according to the guidelines of the National Biobank Network.
IL-33 Inflammatory Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  IL-33 (pg/ml) was measured. The analysis of this inflammatory cytokines was conducted using ELISA (Enzyme-Linked Immunosorbent Assay), with a blood sample obtained according to the guidelines of the National Biobank Network.
HMGB1 Inflammatory Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  HMGB1 (ug/L) was measured. The analysis of this inflammatory cytokines was conducted using ELISA (Enzyme-Linked Immunosorbent Assay), with a blood sample obtained according to the guidelines of the National Biobank Network.
CRP Inflammatory Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  CRP (mg/L) was measured. The analysis of this inflammatory cytokines was conducted using ELISA (Enzyme-Linked Immunosorbent Assay), with a blood sample obtained according to the guidelines of the National Biobank Network.
TNF Inflammatory Profile | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  TNF (pg/ml) was measured. The analysis of this inflammatory cytokines was conducted using ELISA (Enzyme-Linked Immunosorbent Assay), with a blood sample obtained according to the guidelines of the National Biobank Network.

SECONDARY OUTCOMES:
Pittsburg Sleep Quality Index (PSQI) | It was measured before starting treatment and at the end of the treatment, an average of 6 months.
  It is a questionnaire that assess sleep quality and sleep disturbances. It consists of 19 questions that address a wide variety of factors relating to sleep quality, including estimates of sleep duration and latency and of the frequency and severity of sleep-related problems. The 19 items are grouped into seven component scores, each weighted equally on a 0-3 scale. The component scores are summed to give an overall PSQI score between 0 and 21. A higher scores indicates worse sleep quality.
Shoulder mobility | It was measured before starting treatment and at the end of treatment, an average of 6 months.
  Participants' shoulder range of motion will be assessed using an inclinometer. Flexion-extension, abduction-adduction and rotations will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Reina Sofía de Córdoba, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Undecided